CLINICAL TRIAL: NCT00845819
Title: Randomized Phase II Study of Recombinant Human Epidermal Growth Factor (rhEGF) on Oral Mucositis Induced by Intensive Chemotherapy for Hematologic Malignancies
Brief Title: Study of Epidermal Growth Factor on Oral Mucositis Induced by Intensive Chemotherapy for Hematologic Malignancies
Acronym: EGFOM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Principal Investigator, Sung-Soo Yoon, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SNUH-Hema-1001
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Oral Mucositis
Keywords: oral mucositis; intensive chemotherapy; stem cell transplantation; epidermal growth factor
MeSH Terms: conditions — Stomatitis | interventions — Povidone-Iodine; Chlorhexidine; Nystatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EGF (Active Comparator): rhEGF + povidone iodine, chlorhexidine, & nystatin
  Interventions: Drug: rhEGF + povidone iodine, chlorhexidine, & nystatin
- Placebo (Placebo Comparator): Placebo + povidone iodine, chlorhexidine, & nystatin
  Interventions: Drug: Placebo + povidone iodine, chlorhexidine, & nystatin

INTERVENTIONS:
Drug: rhEGF + povidone iodine, chlorhexidine, & nystatin — Topical application of 50 µg/mL rhEGF solution twice daily + oral gargling with povidone iodine (1%), chlorhexidine (0.5%) & nystatin (5,000IU/mL) three times a day.
  Application of drugs begins with start of intensive chemotherapy and ends at the time of recovery from neutropenia (ANC>1000/µL for 3 days) or disappearance of oral mucositis.
  For each application of rhEGF, spray total 6 times at palate, oropharynx, both buccal mucosa, tongue, and gingiva.
  Other Names: Nepidermin; Easyef(R)
  Arms: EGF
Drug: Placebo + povidone iodine, chlorhexidine, & nystatin — Topical application of placebo drug twice daily + oral gargling with povidone iodine (1%), chlorhexidine (0.5%), and nystatin (5,000IU/mL) three times a day.
  Application of drugs begins with start of intensive chemotherapy and ends at the time of recovery from neutropenia (ANC>1000/µL for 3 days) or disappearance of oral mucositis.
  For each application of placebo drug, spray total 6 times at palate, oropharynx, both buccal mucosa, tongue, and gingiva.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine efficacy and toxicity of recombinant human epidermal growth factor (rhEGF) as a preventive drug of oral mucositis during intensive chemotherapy with stem cell transplantation in patients with hematologic malignancies.

DETAILED DESCRIPTION:
Oral mucositis is one of the most common adverse events during chemotherapy and affects quality of life of patients receiving chemotherapy in relation to the dose of drugs. However, there is only one drug (palifermin) approved by the US FDA for the prevention of oral mucositis and the other methods to prevent or treat oral mucositis are just empirical and lack evidences. The results of recent study demonstrated promising efficacy and minimal toxicity of recombinant human epidermal growth factor (rhEGF) as a preventive drug of oral mucositis in head and neck cancer patients undergoing radiotherapy (Wu HG, et al. Cancer 2009;115(16):3699-3708). This clinical trial is a double-blind randomized prospective single-institutional phase II study to evaluate efficacy and toxicity of recombinant human epidermal growth factor (rhEGF) as a preventive drug of oral mucositis during intensive chemotherapy with stem cell transplantation in patients with hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of hematologic malignancies including acute & chronic leukemia, lymphoma, plasma cell dyscrasia, myelodysplastic syndrome, aplastic anemia, etc.
* Patients who are planned to receive high-dose chemotherapy with SCT
* ECOG performance status 0-2
* Informed consent

Exclusion Criteria:

* Patients having previous history of hypersensitivity to this drug or similar drugs
* Patients having oral ulcer or herpes or severe dental disease at the time of inclusion
* Patients received chemotherapy, radiotherapy, or surgery within 3 weeks
* Patients who had finished clinical trials which could affect the results of this trial within 4 weeks or are attending one at the time of inclusion
* Patients having another diseases which have worse prognosis than patients' hematologic malignancy
* Patients with major psychotic disorder or drug/alcohol abuser
* Women who are pregnant or breastfeeding
* Refusal at patients' will
* Inappropriate patients according to the investigators' opinion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2009-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Incidence of oral mucositis of grade 2 or higher (NCI CTCAE 3.0) | Assessed daily during application of study drugs

SECONDARY OUTCOMES:
Adverse events | Assessed daily during application of study drugs
Day of onset and duration of oral mucositis of grade 2 or higher (NCI CTCAE 3.0) | Assessed daily during application of study drugs
Incidence, day of onset, and duration of oral mucositis of grade 3 or higher (NCI CTCAE 3.0) | Assessed daily during application of study drugs
Incidence, day of onset, and duration of oral mucositis of grade 2 or higher (WHO) | Assessed daily during application of study drugs
Incidence, day of onset, and duration of oral mucositis of grade 3 or higher (WHO) | Assessed daily during application of study drugs
Incidence, day of onset, and duration of oral mucositis of grade 4 or higher (WHO) | Assessed daily during application of study drugs
OMDQ (oral mucositis daily questionnaire) score during treatment | Assessed daily during application of study drugs

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Soo Yoon, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Keefe DM, Schubert MM, Elting LS, Sonis ST, Epstein JB, Raber-Durlacher JE, Migliorati CA, McGuire DB, Hutchins RD, Peterson DE; Mucositis Study Section of the Multinational Association of Supportive Care in Cancer and the International Society for Oral Oncology. Updated clinical practice guidelines for the prevention and treatment of mucositis. Cancer. 2007 Mar 1;109(5):820-31. doi: 10.1002/cncr.22484. PMID 17236223
- [Background] Sonis ST, Oster G, Fuchs H, Bellm L, Bradford WZ, Edelsberg J, Hayden V, Eilers J, Epstein JB, LeVeque FG, Miller C, Peterson DE, Schubert MM, Spijkervet FK, Horowitz M. Oral mucositis and the clinical and economic outcomes of hematopoietic stem-cell transplantation. J Clin Oncol. 2001 Apr 15;19(8):2201-5. doi: 10.1200/JCO.2001.19.8.2201. PMID 11304772
- [Background] Brown GL, Curtsinger L 3rd, Brightwell JR, Ackerman DM, Tobin GR, Polk HC Jr, George-Nascimento C, Valenzuela P, Schultz GS. Enhancement of epidermal regeneration by biosynthetic epidermal growth factor. J Exp Med. 1986 May 1;163(5):1319-24. doi: 10.1084/jem.163.5.1319. PMID 3486247
- [Background] Sonis ST, Costa JW Jr, Evitts SM, Lindquist LE, Nicolson M. Effect of epidermal growth factor on ulcerative mucositis in hamsters that receive cancer chemotherapy. Oral Surg Oral Med Oral Pathol. 1992 Dec;74(6):749-55. doi: 10.1016/0030-4220(92)90402-c. PMID 1488231
- [Background] Epstein JB, Gorsky M, Guglietta A, Le N, Sonis ST. The correlation between epidermal growth factor levels in saliva and the severity of oral mucositis during oropharyngeal radiation therapy. Cancer. 2000 Dec 1;89(11):2258-65. doi: 10.1002/1097-0142(20001201)89:113.0.co;2-z. PMID 11147596
- [Background] Hong JP, Lee SW, Song SY, Ahn SD, Shin SS, Choi EK, Kim JH. Recombinant human epidermal growth factor treatment of radiation-induced severe oral mucositis in patients with head and neck malignancies. Eur J Cancer Care (Engl). 2009 Nov;18(6):636-41. doi: 10.1111/j.1365-2354.2008.00971.x. Epub 2009 Apr 23. PMID 19456848
- [Background] Wu HG, Song SY, Kim YS, Oh YT, Lee CG, Keum KC, Ahn YC, Lee SW. Therapeutic effect of recombinant human epidermal growth factor (RhEGF) on mucositis in patients undergoing radiotherapy, with or without chemotherapy, for head and neck cancer: a double-blind placebo-controlled prospective phase 2 multi-institutional clinical trial. Cancer. 2009 Aug 15;115(16):3699-708. doi: 10.1002/cncr.24414. PMID 19514089